CLINICAL TRIAL: NCT01970748
Title: Endoscopic Treatment Versus Propranolol for Primary Prevention of Patients With Hepatocellular Carcinoma and Concomitant Esophageal Varices
Brief Title: Primary Prevention of Patients With Hepatocellular Carcinoma and Concomitant Esophageal Varices
Acronym: P-HCC
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: V101C-016；V102C-094
Record Dates: First submitted 2013-10-22; First posted 2013-10-28 (Estimated); Last update posted 2019-08-30 (Actual); Status verified 2019-08

CONDITIONS: Bleeding Esophageal Varices; Hepatocellular Carcinoma
Keywords: Variceal bleeding; Portal hypertension; Hepatocellular carcinoma; Endoscopic variceal ligation; Non-selective beta-blocker
MeSH Terms: conditions — Carcinoma, Hepatocellular; Hypertension, Portal | interventions — Propranolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Propranolol (Placebo Comparator): Propranolol 10mg BID initially and titrate dosage every week to achieve 25% drop of heart rate (keep heart rate>55 or systemic blood pressure>90mmHg)
  Interventions: Drug: Propranolol
- Esophageal variceal ligation (Active Comparator): Esophageal variceal ligation every 3-4 weeks to achieve variceal eradication under endoscopy. After eradication, follow-up endoscopy every 3 months and variceal ligation again if recurrence.
  Interventions: Procedure: Esophageal variceal ligation

INTERVENTIONS:
Drug: Propranolol — Propranolol 10mg BID initially and titrate dosage every week to achieve 25% drop of heart rate (keep heart rate>55 or systemic blood pressure>90mmHg)
  Other Names: Inderal, Cardolol
  Arms: Propranolol
Procedure: Esophageal variceal ligation — Esophageal variceal ligation every 3-4 weeks to achieve variceal eradication under endoscopy
  Other Names: EVL
  Arms: Esophageal variceal ligation

SUMMARY:
Randomized comparison within the endoscopic esophageal varices ligation versus non-selective beta-blocker in the primary prevention of esophageal variceal bleeding in patients with HCC.

DETAILED DESCRIPTION:
Gastroesophageal variceal bleeding is a major complication of cirrhosis and has high rate of rebleeding and mortality. In these 20 to 30 years, medical advances have significantly improved the prognosis of variceal bleeding. Nevertheless, the mortality of gastroesophageal variceal bleeding is still nearly 20 to 30%.

Hepatocellular carcinoma (HCC) is one of the most common malignancy in Asian, and is also the special group in portal hypertension. Studies in Italy, more than 50% of patients diagnosed with HCC are concomitant with esophageal varices. HCC and portal thrombosis caused by HCC itself are all independent risk factors of gastroesophageal bleeding. Once the bleeding, rebleeding rate is up to 50% even if early use of vasoconstrictor agents and endoscopic therapy, which is generally 2 times in patients with cirrhosis.

According to 2010 Baveno V recommendations, non-selective beta-blockers (NSBB) or endoscopic variceal ligation (EVL) are first choice for primary prevention of first variceal bleeding in cirrhotic patients. However, risk factors of variceal bleeding caused by HCC or cirrhosis are different, and portal hypertension is particularly high in patients with HCC and may be combined with portal vein thrombosis. NSBB sufficient to decreased portal hypertension to prevent variceal bleeding is not clear. In Hepatology 2010, Lebrec claimed that NSBB used for cirrhotic patients with refractory ascites had poor prognosis, the main cause of death were the progression of HCC and sepsis, although the impact of NSBB for HCC patients are not entirely clear, but this issue remind clinicians to careful use of NSBB in these patients. Since NSBB possible adverse effects, the use of EVL to prevent bleeding in patents with HCC is superior to NSBB? These need further study to clarify. So we designed this study to evaluate the feasibility and effectiveness of using EVL or NSBB to prevent first bleeding in patients with HCC concomitant with esophageal varices.

ELIGIBILITY:
Inclusion Criteria:

* Between 20 and 80 years old
* Hepatocellular carcinoma (HCC) associated with esophageal varices
* F2 or F3 esophageal varices (Beppu et al classification)
* Hepatocellular carcinoma (HCC) associated with portal thrombosis

Exclusion Criteria:

* History of esophageal variceal bleeding
* Had received endoscopic variceal ligation (EVL) or endoscopic injection sclerotherapy (EIS)
* Pregnancy, or the patients with other terminal illness (such as other terminal cancers, heart failure, renal failure...)
* Propranolol contraindications (such as atrioventricular block, heart failure, chronic obstructive pulmonary disease, asthma, poorly controlled diabetes, severe peripheral arterial disease...)

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2009-08; Primary Completion 2023-12-25 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Bleeding | 2 years

SECONDARY OUTCOMES:
Complication survival | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Chih Hou, MD, Principal Investigator — Taipei Veterans General Hospital, Taiwan
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Yang TC, Chen WC, Hou MC, Chen PH, Lee PC, Chang CY, Lu HS, Chen YJ, Hsu SJ, Huang HC, Luo JC, Huang YH, Lee FY. Endoscopic variceal ligation versus propranolol for the primary prevention of oesophageal variceal bleeding in patients with hepatocellular carcinoma: an open-label, two-centre, randomised controlled trial. Gut. 2024 Mar 7;73(4):682-690. doi: 10.1136/gutjnl-2023-330419. PMID 38123994